CLINICAL TRIAL: NCT07153952
Title: Evaluation of the Treatment Response and Prognosis of Cervical Adenocarcinoma/Adenosquamous Carcinoma After Radiotherapy Based on Pathologic Characteristics and Multimodal Imaging: a Prospective, Multicenter Trial
Brief Title: RT for Adenocarcinoma/Adenosquamous Carcinoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The First Affiliated Hospital of Xiamen University (Other); Heilongjiang Cancer Hospital (Unknown); Liaoning Cancer Hospital & Institute (Other); Obstetrics and Gynecology Hospital of Zhejiang University (Unknown); Luohe Central Hospital (Unknown)
Responsible Party: Principal Investigator, yanjunfang, Chief Assistant for Department of Radiotherapy, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATTRACT-Pros
Record Dates: First submitted 2025-05-11; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-01

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Radiotherapy
MeSH Terms: interventions — Radiotherapy; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: the local treatment group (Experimental)
  Interventions: Radiation: radiotherapy
- Group B: the systemic treatment group (Active Comparator)
  Interventions: Drug: Systemic treatment

INTERVENTIONS:
Radiation: radiotherapy — The surgical method is determined by the gynecological oncologist, including total hysterectomy, pelvic exenteration, or radical total hysterectomy. The specific surgical choice needs to be comprehensively judged based on the patient's residual tumor location, size, and other complications. Supplementary radiotherapy is mainly image-guided brachytherapy ± external irradiation. The irradiation range and dose must be comprehensively considered based on the location and size of the residual lesions. The best local treatment plan is jointly determined by gynecological oncologists and radiotherapists.
  Arms: Group A: the local treatment group
Drug: Systemic treatment — Systemic treatment regimens include chemotherapy ± targeted therapy ± immunotherapy. According to the NCCN Guidelines (2024.V2), the first-line chemotherapy regimen for persistent, recurrent, or metastatic cervical cancer is preferably carboplatin/paclitaxel and cisplatin/paclitaxel. The addition of immunotherapy can be determined based on the PD-L1 expression level. The specific chemotherapy regimen will be determined by the gynecological oncologist based on the residual tumor site, the number of lesions, and other complications. In addition, if the patient's pathological results indicate HER2 positivity or the genetic test results show PIK3CA mutation, targeted therapy, such as neratinib or apelisimab, can be considered as a second-line regimen after the first-line chemotherapy regimen progresses.
  Arms: Group B: the systemic treatment group

SUMMARY:
This study aims to establish a prospective cohort of locally advanced cervical adenocarcinoma to provide a better way to monitor its efficacy and provide precise treatment. The key problems to be solved are as follows:

1. Establish an observational prospective cohort of locally advanced ADC and randomly divide patients with residual cervical tumors in the primary site after CCRT into the local treatment group (salvage surgery or supplementary radiotherapy) or the systemic treatment group.
2. Collect cervical biopsy tissues before and after CCRT in patients with residual cervical tumors, explore the genomic characteristics, and predict whether they can benefit from targeted/immunotherapy in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of cervical adenocarcinoma;
2. Age 18-80 years old;
3. FIGO 2018 stage IB3-IVA;
4. Karnofsky score≥60 points;
5. Complete blood count, and comprehensive metabolic panel meet the conditions for CCRT;
6. No metal implants in the body, and can perform MRI examination;
7. Willing to participate in this study and provide written informed consent.

Exclusion Criteria:

1. Patients who have received pelvic radiotherapy before;
2. Patients whose target tumors have been treated before (chemotherapy, immunotherapy, surgical treatment, etc.);
3. Allergy to iodine contrast agent;
4. Participating in other clinical studies that may affect the results of this study (determined by the principal investigator);

f) Serious diseases that may significantly affect compliance with clinical trials, such as unstable heart disease, kidney disease, chronic hepatitis, poorly controlled diabetes, and mental illness that require treatment; g) Other situations that the investigator believes are not suitable for participation in this clinical study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Tumor control rate | Tumor control rate among patients with residual cervical tumors in the two groups 3 months after treatment

SECONDARY OUTCOMES:
progression-free survival | 2-year progression-free survival
  The time from randomization to the occurrence of disease recurrence or death from any cause within 2 years was determined based on the time of the first event. If no such event occurred, the time was determined to the last follow-up.
overall survival | 2-year overall survival rate
  The time interval from randomization to death from any cause within 2 years, or if there was no death, to the last follow-up time

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided